CLINICAL TRIAL: NCT04222218
Title: Cerebellar rTMS Theta Burst for Postural Instability in Progressive Supranuclear Palsy: a Double Blind Cross-over Sham-controlled Study Using Wearing Sensors Technology
Brief Title: Cerebellar rTMS Theta Burst for Postural Instability in Progressive Supranuclear Palsy
Acronym: CerTI-PSP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Europea di Ricerca Biomedica Ferb Onlus (Other)
Collaborators: University of Brescia, Neurology Department (Unknown); University of Kiel, Neurogeriatric Department (Unknown)
Responsible Party: Principal Investigator, Andrea Pilotto, parkinson's disease Rehabilitation Centre, Fondazione Europea di Ricerca Biomedica Ferb Onlus
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 191201
Record Dates: First submitted 2019-12-31; First posted 2020-01-09 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Progressive Supranuclear Palsy; Fall; Gait, Rigid; Parkinsonism
Keywords: repetitive Transcranial Magnetic stimulation; cerebellum; wearing sensors; static balance
MeSH Terms: conditions — Supranuclear Palsy, Progressive; Gait Disorders, Neurologic; Parkinsonian Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Each patient received both rTMS and sham cerebellar stimulation in randomized order in two different sessions, separated by at least 2 weeks. In each session, motor tasks, clinical scales and wearing sensor assessments were tested twice in all patients: at baseline (pre-stimulation) and after rTMS (post-stimulation)
Who Masked: Participant, Investigator
Masking Description: The patient and the examiner who administered the clinical scales were blind to the type of rTMS delivered, which was applied by another blinded experimenter.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real Stimulation (Active Comparator): Cerebellar Repetitive theta burst stimulation will be performed using a 3 pulses at 50-Hz repeated at a rate of 5-Hz; 20 trains of 10 bursts given with 8-s intervals for a total of 600 pulses. Intensity of rTMS was set at the 80% of Amplitude of Motor Threshold (RMT) obtained in the left motor cortex for each subject.
  Interventions: Device: repetitive transcranial magnetic stimulation
- Sham Stimulation (Sham Comparator): The rTMS coil stimulation will be applied in the same position of the real stimulation. The Stimulation will be performed like in the real arm with the difference that the coil will be masked and thus will be inactive. The patient will hear the same sound of real stimulation, which will be only functionally inactive but will be completely performed (for the whole time of duration of stimulation)
  Interventions: Device: repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation — Cerebellar repetitive theta Burst stimulation will be performed as detailed in the Real arm description
  Other Names: rTMS; theta Burst, rTMS

SUMMARY:
Objective of the study:

To test the efficacy of theta burst cerebellar stimulation on postural instability in progressive supranuclear palsy using a cross-over design and wearing sensors technology

Design:

Twenty probable PSP patients with no dementia and still able to walk will be recruited for a cross-over sham-controlled study. Each patient will undergo a sham stimulation or a single session of cerebellar theta burst stimulation with a wash out period of at least 14 days.

Each patient will be evaluated before and after stimulation by berg balance tests (BBS), Tinetti scale, PSP-rating scale (PSP-RS), and a battery of gait and movement tests.

Static balance was assessed by 30-seconds-trials in semitandem and tandem positions with eyes open and closed using wearing sensors technology.

DETAILED DESCRIPTION:
Background:

There are no medical effective treatments for progressive supranuclear palsy (PSP). Imaging, neurophysiology and pathology studies suggested cerebellum as possible target of brain stimulation for postural instability using theta Burst repetitive Transcranial magnetic stimulation

Objective of the study:

To test the efficacy of theta burst cerebellar stimulation on postural instability in progressive supranuclear palsy using a cross-over design and wearing sensors technology

Design:

Probable PSP patients able to walk and without dementia/behavioral disturbances will be recruited for a cross-over sham-controlled study. Each patient will undergo a sham stimulation or a single session of cerebellar theta burst stimulation with a wash out period of at least 14 days.

Repetitive cerebellar theta burst stimulation will be performed by Duo-Mag XT100, using a 3 pulses at 50-Hz repeated at a rate of 5-Hz; 20 trains of 10 bursts given with 8-s intervals for a total of 600 pulses. Intensity of rTMS was set at the 80% of Amplitude of Motor Threshold (RMT) obtained in the left motor cortex for each subject.

A sample size of 20 subjects with complete stimulation (2 stimulations per subject, for a total number of stimulation)

Each patient will be evaluated before and after stimulation by berg balance tests (BBS), Tinetti scale, PSP-rating scale (PSP-RS), and a battery of gait and movement tests.

Static balance was assessed by 30-seconds-trials in semitandem and tandem positions with eyes open and closed using wearing sensors technology.

Sensors assessment:

The following parameters will be evaluated before and after stimulation (real vs sham): The parameter i) TIME, defined as time without falling ii) The parameter "surface", defined as the sway area iii) Velocity describes the mean velocity of the compensatory movements given in mm/s. iv) Acceleration described as root mean square (RMS), v) Jerk, the time derivate of acceleration, quantifies smoothness of the compensatory movements given in mG/s.

ELIGIBILITY:
Inclusion Criteria:

* probable PSP diagnosis
* ability to stand alone without support for at least 5 seconds
* ability to walk without aid for at least three meters

Exclusion Criteria:

* dementia or behavioral alterations
* contraindications of stimulation

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Short Physical Performance Battery, total time (SPPB) | Changes from Baseline to immediately after stimulation
  The short Physical performance battery included a walking test at convenient speed, a chair-rise test at convenient speed and tests of static balance including feet together, semi-tandem and tandem stance)
Timed up and Go tests, total time (TUG) | Changes from Baseline to immediately after stimulation
  The time of performance of two timed up and go test ( one starting with the right foot, one starting with the left foot) will be assessed
Static Balance tests, total time | Changes from Baseline to immediately after stimulation
  The assessment of static balance will include four tasks, in which the patient has to stand alone and maintain the position in different conditions for up to 30 seconds: tandem and semitandem positions with eyes closed and eyes open, respectively.
  The time of performance without falling will be assessed.
Tinetti Balance test (TBT) | Changes from Baseline to immediately after stimulation
  Assessment of postural instability (0-28, higher scores indicate better performances)
Static Balance- area of sway | Changes from Baseline to immediately after stimulation
  The area of sway during the postural instability tasks will be assessed (unit of measure mm2)

SECONDARY OUTCOMES:
PSP rating scale (PSP-RS) | Changes from Baseline to immediately after stimulation
  Assessment of postural instability and disability of patients (scores ranging from 0 to 100, lower scores indicate less disability)
Static Balance: wearable sensor analyses - velocity | Changes from Baseline to immediately after stimulation
  the velocity of sway will be assessed during the postural instability tasks (unit of measure (mm/s)
Static Balance: wearable sensor analyses - acceleration | Changes from Baseline to immediately after stimulation
  the acceleration of sway will be assessed during the postural instability tasks (unit of measure mm2/s)
Static Balance: wearable sensor analyses - jerk | Changes from Baseline to immediately after stimulation
  The time-derived of acceleration of sway will be assessed during the postural instability tasks (unit of measure mm3/s)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Pilotto, MD, Principal Investigator — Università degli Studi di Brescia
Locations (1):
- Parkinson's disease Rehabilitation Centre - FERB ONLUS, Trescore Balneario, Italy

IPD SHARING:
Plan to Share IPD: Yes
The whole project will be published in medical journal
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: In the publication, within the next year
Access Criteria: on-line availability